CLINICAL TRIAL: NCT02211326
Title: Pharmacogenetic Algorithm of Response to Warfarin During Initial Anticoagulation in Chinese Elderly Patients
Brief Title: Genotype-guided Warfarin Individualized Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XY3-WARF1405A01; ChiCTR-TRC-14004757 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2014-08-06; First posted 2014-08-07 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Atrial Fibrillation; Deep Venous Thrombosis
Keywords: AF or DVT; Age Over 18 Years, Acquired
MeSH Terms: conditions — Atrial Fibrillation; Venous Thrombosis | interventions — Warfarin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- genotype-guided group (Experimental): Interventions：on day1~day3, patients received dose according to IWPC formula (PGx-1) included clinical variables and genotype data for VKORC1, CYP2C9*1, CYP2C9*2, and CYP2C9*3; on day4~day7, patients received dose according to Lenzini formula consisted of clinical variables, VKORC1, CYP2C9*2, CYP2C9*3 and previous INR and dosing information (PGx-2); and on day8, the clinicians adjusted the dose according to observed INR.The overall follow-up period is 12 weeks.
  Interventions: Behavioral: Genotype-guided dosing algorithm for warfarin
- control group (Active Comparator): Interventions：on day1~day3, patients were given initial dose (2.25mg); and starting from day4, the clinicians began to adjust the dose for patients according to observed INR.The overall follow-up period is 12 weeks.
  Interventions: Behavioral: Standard initiation dose for warfarin

INTERVENTIONS:
Behavioral: Genotype-guided dosing algorithm for warfarin — Intervention：initial dosing of warfarin for the first 3 days of treatment will be determined by IWPC( International Warfarin Pharmacogenetics Consortium) algorithm (PG-1),a second dose adjustment will be made after 3 doses of warfarin using a dose revision algorithm (PG-2) that combined INR values,the dose will be adjusted depending on the measurements of INR values after 7 days.The overall follow-up period is 12 weeks.
  Arms: genotype-guided group
Behavioral: Standard initiation dose for warfarin — Intervention：initial dosing of warfarin for the first 3 days of treatment will be determined by standard initiation dose. Following this initiation dose of warfarin,the dose will be adjusted depending on the measurements of INR values after 3 days.The overall follow-up period is 12 weeks.
  Arms: control group

SUMMARY:
The purpose of this study is to determine whether the international pharmacogenetic algorithm is better than the standard initiation dosing and whether the two algorithms are suitable for Chinese elderly patients.

DETAILED DESCRIPTION:
The study protocol is a multicenter, randomized, patient-blinded and controlled trial, comparing two approaches among 864 enrolled AF(atrial fibrillation) or DVT(deep venous thrombosis) patients for guiding warfarin initial anticoagulation in Chinese elderly patients: the intervention group using the algorithm of International Warfarin Pharmacogenetic Consortium and its dose revision, and the control group using a standard initiation dose (2.25 mg).The study hypothesis is that the intervention group relative to the control group will increase the percentage of time in therapeutic INR (international normalized ratio) range during the first 3 months.This trial is the first prospective large-scale randomized controlled trial for elders in China. It is of great significance for promoting special crowd individualization of anticoagulants at home and abroad.

ELIGIBILITY:
Inclusion criteria：1) Chinese male or female aged ≥18 years; 2) Requiring at least 12-week warfarin therapy as judged by clinicians; 3) Subjects with DVT/AF and a post-therapy target INR of 1.5-2.5; 4) Capable of providing written informed consent; 5) Capable of maintaining excellent communications with investigators and completing trial in accordance with trial stipulations.

Exclusion criteria：1) Subjects previously taking warfarin; 2) Known genotypes of CYP2C9 or/and VKORC1; 3) Subjects receiving or expecting to receive other therapies or other anticoagulants; 4) Subjects with contraindications for warfarin; 5) Subjects with severe cognitive dysfunctions; 6) Baseline INR ≥1.5; 7) Subjects with drug or alcohol dependence within the last 12 months; 8) Subjects receiving blood transfusion or bone marrow transplantation within the last 2 weeks; 9) Planning to receive invasive examinations (except for standard endoscopy) with a hemorrhagic tendency or undergoing surgery during trial.10) Prior to randomization, subjects receiving any trial drug or device within the last 3 months or planning to receive such an investigational therapy during trial; 11) Subjects with the following diagnoses or conditions: active malignant carcinomas (diagnosed within the last 5 years), but excluding adequately-treated non-melanoma skin cancer or other non-invasive or in situ cancer (e.g. cervical cancer in situ); anti-neoplastic therapy within the last 5 years (medication, radiotherapy or/and surgery); overt active disease or infection; life expectancy <6 months; 12）Other clinical reasons for unsuitable recruitment as judged by clinicians.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2017-01-16 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
%TTR | 12 weeks
  percentage of time in the therapeutic INR (%TTR) of INR 2-3 (<60 years old) or 1.5-2.5 (≥ 60 years old) within 12 weeks

SECONDARY OUTCOMES:
the time to reach therapeutic INR | 12 weeks
  the time to reach therapeutic INR
the time to reach stable warfarin dose which defined as the dose to achieve INR within ±0.1 of therapeutic range at Day 8 post-dose | 12 weeks
  the time to reach stable warfarin dose which defined as the dose to achieve INR within ±0.1 of therapeutic range at Day 8 post-dose
The number of adjustment units in the dose of warfarin (with 0.375 mg (1/8 tablet) as a unit); Incidence of INR ≥ 4 | 12 weeks
  The number of adjustment units in the dose of warfarin (with 0.375 mg (1/8 tablet) as a unit); Incidence of INR ≥ 4

OTHER OUTCOMES:
the number of additional clinic visits | 12 weeks
  the number of additional clinic visits

CONTACTS AND LOCATIONS:
Overall Officials: GuoPing Yang, professor, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (15):
- China (15):
  - The People's Hospital of Hunan Province, Changsha, Hunan
  - The Central Hospital of Changsha, Changsha, Hunan
  - The Fourth Hospital of Changsha, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Hospital of Changsha, Changsha, Hunan
  - The Xiangya Hospital of Central South University, Changsha, Hunan
  - The First People's Hospital of Chenzhou, Chenzhou, Hunan
  - The First Affiliated Hospital of Nanhua university, Hengyang, Hunan
  - The Second Affiliated Hospital of Nanhua university, Hengyang, Hunan
  - The Central Hospital of Loudi, Loudi, Hunan
  - The Central Hospital of Shaoyang, Shaoyang, Hunan
  - The First People's Hospital of Shaoyang, Shaoyang, Hunan
  - The Central Hospital of Xiangtan, Xiangtan, Hunan
  - The First People's Hospital of Xiangtan, Xiangtan, Hunan
  - The Central Hospital of Yiyang, Yiyang, Hunan

REFERENCES:
- [Background] Eikelboom JW, Connolly SJ, Brueckmann M, Granger CB, Kappetein AP, Mack MJ, Blatchford J, Devenny K, Friedman J, Guiver K, Harper R, Khder Y, Lobmeyer MT, Maas H, Voigt JU, Simoons ML, Van de Werf F; RE-ALIGN Investigators. Dabigatran versus warfarin in patients with mechanical heart valves. N Engl J Med. 2013 Sep 26;369(13):1206-14. doi: 10.1056/NEJMoa1300615. Epub 2013 Aug 31. PMID 23991661
- [Background] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957
- [Background] Giugliano RP, Ruff CT, Braunwald E, Murphy SA, Wiviott SD, Halperin JL, Waldo AL, Ezekowitz MD, Weitz JI, Spinar J, Ruzyllo W, Ruda M, Koretsune Y, Betcher J, Shi M, Grip LT, Patel SP, Patel I, Hanyok JJ, Mercuri M, Antman EM; ENGAGE AF-TIMI 48 Investigators. Edoxaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2013 Nov 28;369(22):2093-104. doi: 10.1056/NEJMoa1310907. Epub 2013 Nov 19. PMID 24251359
- [Background] Arepally GM, Ortel TL. Changing practice of anticoagulation: will target-specific anticoagulants replace warfarin? Annu Rev Med. 2015;66:241-53. doi: 10.1146/annurev-med-051113-024633. PMID 25587651
- [Background] Healey JS, Oldgren J, Ezekowitz M, Zhu J, Pais P, Wang J, Commerford P, Jansky P, Avezum A, Sigamani A, Damasceno A, Reilly P, Grinvalds A, Nakamya J, Aje A, Almahmeed W, Moriarty A, Wallentin L, Yusuf S, Connolly SJ; RE-LY Atrial Fibrillation Registry and Cohort Study Investigators. Occurrence of death and stroke in patients in 47 countries 1 year after presenting with atrial fibrillation: a cohort study. Lancet. 2016 Sep 17;388(10050):1161-9. doi: 10.1016/S0140-6736(16)30968-0. Epub 2016 Aug 8. PMID 27515684
- [Derived] Kuang Y, Liu Y, Pei Q, Ning X, Zou Y, Liu L, Song L, Guo C, Sun Y, Deng K, Zou C, Cao D, Cui Y, Wu C, Yang G. Long Short-Term Memory Network for Development and Simulation of Warfarin Dosing Model Based on Time Series Anticoagulant Data. Front Cardiovasc Med. 2022 May 11;9:881111. doi: 10.3389/fcvm.2022.881111. eCollection 2022. PMID 35647078
- [Derived] Ning X, Kuang Y, Yang G, Xie J, Miao D, Guo C, Huang Z. Influence of renal insufficiency on anticoagulant effects and safety of warfarin in Chinese patients: analysis from a randomized controlled trial. Naunyn Schmiedebergs Arch Pharmacol. 2021 Jun;394(6):1275-1283. doi: 10.1007/s00210-020-02037-3. Epub 2021 Jan 6. PMID 33404689
- [Derived] Guo C, Kuang Y, Zhou H, Yuan H, Pei Q, Li J, Jiang W, Ng CM, Chen X, Huo Y, Cui Y, Wang X, Yu J, Sun X, Yu W, Chen P, Miao D, Liu W, Yu Z, Ouyang Z, Shi X, Lv C, Peng Z, Xiong G, Zeng G, Zeng J, Dai H, Peng J, Zhang Y, Xu F, Wu J, Chen X, Gong H, Yang Z, Wu X, Fang Q, Yang L, Li H, Tan H, Huang Z, Tang X, Yang Q, Tu S, Wang X, Xiang Y, Huang J, Wang X, Cai J, Jiang S, Huang L, Peng J, Gong L, Zou C, Yang G. Genotype-Guided Dosing of Warfarin in Chinese Adults: A Multicenter Randomized Clinical Trial. Circ Genom Precis Med. 2020 Aug;13(4):e002602. doi: 10.1161/CIRCGEN.119.002602. Epub 2020 Jun 8. PMID 32510984